CLINICAL TRIAL: NCT06415981
Title: Single Center Proof-of-Concept Study to Determine the Flow Changes When Stimulating Two Neural Targets for the Treatment of Obstructive Sleep Apnea
Brief Title: Proof-of-Concept Study to Determine the Flow Changes When Stimulating Two Neural Targets for the Treatment of Obstructive Sleep Apnea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Invicta Medical Inc. (Industry)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM-003
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive; Sleep Disorder; Sleep Apnea Syndromes
Keywords: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hypoglossal nerve and/or Ansa Cervicalis stimulation (Experimental)
  Interventions: Device: Hypoglossal nerve and/or Ansa Cervicalis stimulation

INTERVENTIONS:
Device: Hypoglossal nerve and/or Ansa Cervicalis stimulation — Device stimulation of the hypoglossal nerve and/or Ansa Cervicalis

SUMMARY:
This proof-of-concept study will evaluate the impact of surgically placing and stimulating the hypoglossal nerve and/or a second neural target Ansa Cervicalis, with a set of off-the-shelf electrode arrays.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years not under guardianship, under curatorship or under judicial protection.
* Body Mass Index (BMI) < 35 kg/m2.
* Subject suffers from OSA (15 < AHI < 80) documented by a sleep study performed during the past 36 months.
* Subject must be eligible for a diagnostic or surgical procedure.
* Written informed consent obtained from the patient prior to performing any study specific procedure.
* Willing and capable to comply with all study requirements, including specific lifestyle considerations, evaluation procedures and questionnaires for the whole duration of the trial.

Exclusion Criteria:

* Major anatomical or functional abnormalities that would impair the ability of the electrode arrays to be positioned
* Significant comorbidities that contraindicate surgery or general anesthesia
* Significant tongue weakness
* Any other chronic medical illness or condition that contraindicates a surgical procedure or general anesthesia in the judgment of the investigator.
* Prior surgery or treatments that could compromise the placement and effectiveness of the electrode array systems:
* Airway cancer surgery or radiation,
* Mandible or maxilla surgery in the previous 3 years (not counting dental treatments),
* Other upper airway surgery to remove obstructions related to OSA in the previous 3 months (e.g., uvulopalatopharyngoplasty (UPPP), tonsillectomy, nasal airway surgery),
* Prior hypoglossal nerve stimulation device implantation.
* Currently pregnant, or breastfeeding during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with changes in cross-sectional area airway opening during target stimulation | Day 0
  Assessment of patients with changes in acute cross-sectional area airway opening measured in cm2 under nasoendoscopy when stimulating two neural targets (the HGN and AC). Video imaging and physician interpretation of nasoendoscopic images will be used to review outcome measures.
Assessment of changes in airflow outcomes | Day 0
  Assessment of acute changes in airflow when stimulating the HGN in combination with the AC during a flow limited event (hypopnea or apnea).

SECONDARY OUTCOMES:
Number of participant adverse events observed during the study | Day 30
  To evaluate and report all observed participant adverse events observed during study.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No